CLINICAL TRIAL: NCT07195916
Title: A Phase 1, Open-Label, Multicenter Study of INCA036873 in Participants With Advanced Solid Tumors and Hematological Malignancies
Brief Title: A Study to Evaluate INCA036873 in Participants With Advanced Solid Tumors and Hematological Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INCA036873-101; 2025-523130-11-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2025-09-19; First posted 2025-09-29 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Solid Tumors; Hematologic Malignancies
Keywords: Advanced solid tumors; Metastatic solid tumors; Clear cell renal cell carcinoma (ccRCC); Diffuse large B-cell lymphoma (DLBCL); High-grade B-cell lymphoma (HGBCL); Peripheral T-cell lymphoma (PTCL, incl. ALCL); Cutaneous T-cell lymphoma (CTCL, incl. MF and SS); Non-Hodgkin lymphoma (NHL); CD70; Bispecific antibody; Immunotherapy; T-cell engager
MeSH Terms: conditions — Hematologic Neoplasms; Carcinoma, Renal Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell, Cutaneous; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1a Dose Escalation (Experimental): INCA036873 will be administered at the protocol defined dose.
  Interventions: Drug: INCA036873
- Part 1b Dose Expansion (Experimental): INCA036873 will be administered at the protocol defined dose.
  Interventions: Drug: INCA036873
- Part 1c Pharmacodynamic Cohort (Experimental): INCA036873 will be administered at the protocol defined dose.
  Interventions: Drug: INCA036873

INTERVENTIONS:
Drug: INCA036873 — Intravenously (IV)

SUMMARY:
A study to evaluate the safety and tolerability of INCA036873 in participants with advanced solid tumors and hematological malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* ECOG performance status of 0 or 1.
* Histologically confirmed:

  * Clear cell renal cell carcinoma (ccRCC).
  * Diffuse large B-cell lymphoma (DLBCL, NOS).
  * High-grade B-cell lymphoma (HGBCL).
  * Peripheral T-cell lymphoma (PTCL, incl. NOS and ALCL).
  * Cutaneous T-cell lymphoma (CTCL, incl. MF or SS ≥Stage IIB with B0/B1 blood involvement).
* Disease progression, relapse, or refractory to prior therapy:

  * ccRCC: ≥1 prior line incl. ICI + TKI.
  * DLBCL/HGBCL: ≥2 prior lines incl. immunochemotherapy and salvage.
  * PTCL/CTCL: ≥1 prior systemic therapy.
* Measurable disease by RECIST v1.1 (ccRCC), Lugano 2014 (lymphomas), or ISCL/USCLC/EORTC (CTCL).
* Tumor tissue available for central testing.

Exclusion Criteria:

* Untreated or progressive CNS disease unless previously treated and stable.
* Other active invasive malignancy within 2 years (except certain low-risk cancers).
* Prior CD70-targeting therapy, including CAR T.
* ASCT or CAR T ≤12 weeks before enrollment; prior organ or allogeneic transplant.
* Unresolved ≥Grade 2 toxicity from prior therapy (with exceptions).
* Primary immunodeficiency or active autoimmune disease requiring immunosuppression.
* Active HBV, HCV, HIV, or other chronic infections requiring systemic therapy.
* Pregnancy, breastfeeding, or unwillingness to use effective contraception.

Other protocol-defined Inclusion/Exclusion Criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2026-01-08 (Actual); Primary Completion 2028-08-18 (Estimated); Study Completion 2028-08-18 (Estimated)

PRIMARY OUTCOMES:
Part 1A : Occurrence of Dose Limiting Toxicities (DLTs) | Up to Day 28
  Toxicities occurring during the first study drug infusion and continues through 28 days as defined in the protocol. DLTs will be assessed for severity by the investigator using CTCAE v5.0 criteria.
Number of Participants With Treatment Emergent Adverse Events (TEAEs) | Up to approximately 2 years and 90 days
  TEAE is any Adverse Event (AE) either reported for the first time or worsening of a pre-existing event after first dose of study drug.

SECONDARY OUTCOMES:
Pharmacokinetics Parameter: Cmax of INCA036873 | Up to approximately 2 years and 90 days
  Defined as maximum observed plasma concentration of INCA036873.
Pharmacokinetics Parameter: Tmax of INCA036873 | Up to approximately 2 years and 90 days
  Defined as the time to reach the maximum plasma concentration of INCA036873.
Pharmacokinetics Parameter: Cmin of INCA036873 | Up to approximately 2 years and 90 days
  Defined as the minimum observed plasma concentration of INCA036873.
Pharmacokinetics Parameter: AUC(0-t) of INCA036873 | Up to approximately 2 years and 90 days
  Defined as the area under the concentration-time curve up to the last measurable concentration of INCA036873.
Pharmacokinetics Parameter: AUC 0-∞ of INCA036873 | Up to approximately 2 years and 90 days
  Defined as the area under the concentration-time curve from 0 to infinity of INCA036873.
Pharmacokinetics Parameter: CL of INCA036873 | Up to approximately 2 years and 90 days
  Defined as the apparent oral dose clearance of INCA036873.
Pharmacokinetics Parameter: Vz of INCA036873 | Up to approximately 2 years and 90 days
  Defined as the apparent oral dose volume of distribution of INCA036873.
Pharmacokinetics Parameter: t1/2 of INCA036873 | Up to approximately 2 years and 90 days
  Defined as the apparent terminal phase disposition half-life of INCA036873.
Objective response | Up to approximately 2 years
  Defined as a Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR), as assessed by the investigator.
Disease control | Up to approximately 2 years
  Defined as a BOR of CR, PR, or Stable Disease (SD), as assessed by the investigator.
Duration of Response (DOR) | Up to approximately 2 years
  Defined as the time from the earliest date of a documented objective response (CR or PR) to the earliest date of disease progression (per investigator assessment using the appropriate criteria) or death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Study Monitor, Study Director — Incyte Corporation
Locations (22):
- United States (8):
  - City of Hope Medical Center, Duarte, California
  - University of California San Diego Medical Center, Moores Cancer Center, La Jolla, California
  - University of Michigan, Ann Arbor, Michigan
  - The University of Nebraska Medical Center, Omaha, Nebraska
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Scri Oncology Partners, Nashville, Tennessee
  - Vanderbilt Medical Center, Nashville, Tennessee
  - Md Anderson Cancer Center, Houston, Texas
- Australia (4):
  - Macquarie University Hospital, Sydney, New South Wales
  - Princess Alexandra Hospital Australia, Woolloongabba, Queensland
  - Cancer Research Sa, Adelaide, South Australia
  - Peter Maccallum Cancer Centre-Royal Melbourne Hospital, Melbourne, Victoria
- Belgium (4):
  - Cliniques Universitaires Ucl Saint-Luc, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Universitair Ziekenhuis Gent (Uz Gent), Ghent
  - Universitair Ziekenhuis Leuven, Leuven
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet Uni of Hospital of Copenhagen, Copenhagen
- Italy (4):
  - Aou Policlinico S. Orsola-Malpighi, Bologna
  - Fondazione Irccs Istituto Nazionale Dei Tumori, Milan
  - Policlinico Universitario Agostino Gemelli Universita Cattolica Del Sacro Cuore, Rome
  - Centro Ricerche Cliniche Di Verona, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study to Evaluate INCA036873 in Participants With Advanced Solid Tumors and Hematological Malignancies — https://incyteclinicaltrials.com/studies/nct07195916